CLINICAL TRIAL: NCT00887224
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized Withdrawal, Parallel Group Study To Evaluate The Efficacy And Safety Of 50 mg/Day Of DVS SR In Adult Outpatients With Major Depressive Disorder
Brief Title: Relapse Prevention Study Of Desvenlafaxine Succinate Sustained Release In Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3151A1-3360; B2061004
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desvenlafaxine succinate sustained release 50 mg (Experimental)
  Interventions: Drug: Desvenlafaxine succinate sustained release 50 mg; Drug: Desvenlafaxine succinate sustained release 25 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine succinate sustained release 50 mg — 50 mg tablet, once daily. 5 months open-label duration for all enrolled subjects; additional 6 months double-blind duration for randomized subjects assigned to this arm.
  Other Names: Pristiq
  Arms: Desvenlafaxine succinate sustained release 50 mg
Drug: Desvenlafaxine succinate sustained release 25 mg — 25 mg tablet for taper, once daily for 1 week
  Other Names: Pristiq
  Arms: Desvenlafaxine succinate sustained release 50 mg
Drug: Placebo — Matching placebo tablet, once daily. 6 months double-blind duration for randomized subjects assigned to placebo.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to compare the long-term efficacy and safety of desvenlafaxine succinate sustained release versus placebo in adults with Major Depressive Disorder, using a randomized withdrawal design. Randomized withdrawal means that after receiving desvenlafaxine succinate sustained release for a predetermined period of time, subjects will be selected by chance to either continue receiving the study drug or to be withdrawn from the study drug and receive placebo for the remainder of their participation in the trial. Subjects will not know to which group they have been assigned.

The study consists of an up to 14-day screening period followed by an 8-week open-label period in which subjects will knowingly receive 50 mg/day of desvenlafaxine succinate sustained release. Subjects who do not respond to treatment, demonstrating no significant change in their depressive symptoms, will be withdrawn from participation at the end of this period. Responding subjects will receive an additional 3 months of open-label desvenlafaxine succinate sustained release at the same dose. Subjects with stable response to treatment at the conclusion of this 3 month period will be randomized to either desvenlafaxine succinate sustained release at 50 mg/day or placebo in a blinded manner for an additional 6 months or until symptoms of depression return. Following discontinuation at any point after enrollment in the study, subjects will receive two weeks of follow-up monitoring, including one week of blinded taper with 25 mg/day of desvenlafaxine succinate sustained release treatment for any subjects who have been taking desvenlafaxine succinate sustained release prior to discontinuation. Subjects assigned to placebo will receive a blinded placebo taper. Following taper, subjects will be evaluated for one additional week to monitor safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult, outpatient with primary diagnosis of Major Depressive Disorder (depressive symptoms for at least 30 days prior to screening)
* Hamilton Psychiatric Rating Scale for Depression (HAM-D 17) total score of >= 20
* Clinical Global Impressions Scale-Severity (CGI-S) score of >= 4.

Exclusion Criteria:

* Significant risk of suicide as assessed by clinician judgment, HAM-D17 and Columbia Suicide-Severity Rating Scale scores.
* Past treatment with desvenlafaxine succinate sustained release.
* Other eligibility criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (80):
- United States (19):
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Smyrna, Georgia
  - Pfizer Investigational Site, Hoffman Estates, Illinois
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington
- Canada (11):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Medicine Hat, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Bathurst, New Brunswick
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Gatineau, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Pfizer Investigational Site, Santiago, Chile, Chile
- Colombia (4):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Bucamaranga, Santander Department
- Croatia (2):
  - Pfizer Investigational Site, Rijeka
  - Pfizer Investigational Site, Zagreb
- Estonia (4):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
  - Pfizer Investigational Site, Võru
  - Pfizer Investigational Site, Vöru
- Finland (7):
  - Pfizer Investigational Site, Espoo
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Joensuu
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Seinäjoki
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- France (6):
  - Pfizer Investigational Site, Douai, France
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Dole
  - Pfizer Investigational Site, Douai
  - Pfizer Investigational Site, Orvault
  - Pfizer Investigational Site, Rennes
- Latvia (4):
  - Pfizer Investigational Site, Strenči, Latvia
  - Pfizer Investigational Site, Liepāja
  - Pfizer Investigational Site, Sigulda
  - Pfizer Investigational Site, Strenči
- Lithuania (3):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilius
  - Pfizer Investigational Site, Vilnius
- Poland (6):
  - Pfizer Investigational Site, Skorzewo, Poznan
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Tuszyn
  - Pfizer Investigational Site, Wroclaw
  - Pfizer Investigational Site, Żuromin
- Romania (4):
  - Pfizer Investigational Site, Brasov, Brașov County
  - Pfizer Investigational Site, Craiova, Dolj
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Cluj-Napoca
- Slovakia (6):
  - Pfizer Investigational Site, Bojnice
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Liptovský Mikuláš
  - Pfizer Investigational Site, Michalovce
  - Pfizer Investigational Site, Rimavská Sobota
  - Pfizer Investigational Site, Trenčín
- South Africa (3):
  - Pfizer Investigational Site, Cape Town, Western Cape
  - Pfizer Investigational Site, Durban
  - Pfizer Investigational Site, Paarl

REFERENCES:
- [Derived] Boyer P, Vialet C, Hwang E, Tourian KA. Efficacy of Desvenlafaxine 50 mg/d Versus Placebo in the Long-Term Treatment of Major Depressive Disorder: A Randomized, Double-Blind Trial. Prim Care Companion CNS Disord. 2015 Aug 27;17(4):10.4088/PCC.14m01711. doi: 10.4088/PCC.14m01711. eCollection 2015. PMID 26693033
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. An Analysis of Relapse Rates and Predictors of Relapse in 2 Randomized, Placebo-Controlled Trials of Desvenlafaxine for Major Depressive Disorder. Prim Care Companion CNS Disord. 2015 Feb 26;17(1):10.4088/PCC.14m01681. doi: 10.4088/PCC.14m01681. eCollection 2015. PMID 26137355
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Rosenthal JZ, Boyer P, Vialet C, Hwang E, Tourian KA. Efficacy and safety of desvenlafaxine 50 mg/d for prevention of relapse in major depressive disorder:a randomized controlled trial. J Clin Psychiatry. 2013 Feb;74(2):158-66. doi: 10.4088/JCP.12m07974. PMID 23473348
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-3360&StudyName=Relapse%20Prevention%20Study%20Of%20Desvenlafaxine%20Succinate%20Sustained%20Release%20In%20Outpatients%20With%20Major%20Depressive%20Disorder

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1072 participants were screened, 874 were enrolled into Desvenlafaxine succinate sustained release (DVS SR) open-label 8-week response phase; 659 entered into 12-week open label stability phase. After 20 weeks of open-label treatment 548 subjects were randomized to the 6-month double-blind phase to receive either placebo or to continue with DVS SR.
Groups:
- DVS SR 50 mg (Open-label Phase): Desvenlafaxine succinate sustained release (DVS SR) 50 milligrams (mg) by mouth (PO) once daily (QD) for 20 weeks (Days 1 to 140). This included an 8-week response phase and for responders at Week 8, a 12-week stability phase. Participants who concluded open-label study or discontinued treatment received DVS SR 25 mg PO QD for 7-day taper period (All Enrolled Population).
- Placebo (Double-blind Phase): Placebo matching DVS SR 50 mg and DVS SR 25 mg PO QD Days 141 to 147, then placebo matching DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with placebo matching DVS SR 25 mg PO QD (All Randomized Population).
- DVS SR 50 mg (Double-blind Phase): DVS SR 50 mg and placebo matching DVS SR 25 mg PO QD Days 141 to 147; DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with DVS SR 25 mg PO QD (All Randomized Population).
Period: Open-label Response (OLR) Phase
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase)
Started | 874 | 0 | 0
Completed | 752 | 0 | 0
Not Completed | 122 | 0 | 0
Not completed — Adverse Event | 46 | 0 | 0
Not completed — Failed to return | 6 | 0 | 0
Not completed — Lack of Efficacy | 26 | 0 | 0
Not completed — Lost to Follow-up | 16 | 0 | 0
Not completed — Other | 1 | 0 | 0
Not completed — Protocol Violation | 12 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 0 | 0
Period: Between OLR and OLS Phases
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase)
Started | 752 | 0 | 0
Completed | 659 | 0 | 0
Not Completed | 93 | 0 | 0
Period: Open-label Stability (OLS) Phase
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase)
Started | 659 | 0 | 0
Completed | 576 | 0 | 0
Not Completed | 83 | 0 | 0
Not completed — Adverse Event | 22 | 0 | 0
Not completed — Failed to return | 3 | 0 | 0
Not completed — Lack of Efficacy | 16 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0
Not completed — Other | 1 | 0 | 0
Not completed — Protocol Violation | 13 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 0 | 0
Period: Between OLS and DB Phases
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase)
Started | 576 | 0 | 0
Completed | 548 | 0 | 0
Not Completed | 28 | 0 | 0
Period: OL Taper Phase / OL Follow Up
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase)
Started | 307 (Could have entered 7-day taper period at any time during either the OLR phase or OLS phase.) | 0 | 0
Discontinued Open-label Taper | 144 (Could have discontinued at any time during OL taper phase or OL Follow-up (7 days after last dose).) | 0 | 0
Completed | 163 | 0 | 0
Not Completed | 144 | 0 | 0
Not completed — Adverse Event | 28 | 0 | 0
Not completed — Failed to return | 17 | 0 | 0
Not completed — Physician Decision | 10 | 0 | 0
Not completed — Lost to Follow-up | 8 | 0 | 0
Not completed — Other | 30 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Withdrawal by Subject | 48 | 0 | 0
Period: Double-blind (DB) Phase
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase)
Started | 0 | 276 (2 participants randomized in error to DB, then entered OL Taper; counted in OL Taper and DB phases.) | 272
Completed | 0 | 176 | 210
Not Completed | 0 | 100 | 62
Not completed — Adverse Event | 0 | 7 | 2
Not completed — Failed to return | 0 | 2 | 2
Not completed — Lack of Efficacy | 0 | 67 | 33
Not completed — Lost to Follow-up | 0 | 8 | 8
Not completed — Other | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 8 | 5
Not completed — Withdrawal by Subject | 0 | 6 | 12
Period: DB Taper Phase / Post Study Follow Up
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase)
Started | 0 | 267 (Double-blind participants (DBp) could have entered 7-day taper period at any time during DB phase.) | 265
Did Not Enter DB Taper | 0 | 9 | 7
Discontinued DB Taper | 0 | 41 (DBp could have discontinued at anytime during DB taper period or Follow-up (7 days after last dose).) | 30
Completed | 0 | 226 | 235
Not Completed | 0 | 41 | 30
Not completed — Adverse Event | 0 | 5 | 0
Not completed — Failed to return | 0 | 5 | 4
Not completed — Physician Decision | 0 | 6 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Other | 0 | 11 | 12
Not completed — Protocol Violation | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- DVS SR 50 mg (Open-label Phase): DVS SR 50 mg PO QD for 20 weeks (Days 1 to 140). This included an 8-week response phase and for responders at Week 8, a 12-week stability phase. Participants who concluded open-label study or discontinued treatment received DVS SR 25 mg PO QD for 7-day taper period (All Enrolled Population).
- Placebo (Double-blind Phase): Eligible participants from OL Phase were randomized in a 1:1 ratio to either Placebo or DVS SR in the DB Phase.
  Placebo matching DVS SR 50 mg and DVS SR 25 mg PO QD Days 141 to 147, then placebo matching DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with placebo matching DVS SR 25 mg PO QD (All Randomized Population).
- DVS SR 50 mg (Double-blind Phase): Eligible participants from OL Phase were randomized in a 1:1 ratio to either Placebo or DVS SR in the DB Phase.
  DVS SR 50 mg and placebo matching DVS SR 25 mg PO QD Days 141 to 147; DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with DVS SR 25 mg PO QD (All Randomized Population).
- Total: Total of all reporting groups
Arm/Group | DVS SR 50 mg (Open-label Phase) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase) | Total
Number analyzed (Participants) | 874 | 276 | 272 | 1422
Age, Continuous [Mean (Standard Deviation); unit: years] — OL Baseline All Enrolled Population
  years | 44.98 (13.25) | NA (NA) — Baseline Age reported for participants entering the Open-label phase at study start. | NA (NA) — Baseline Age reported for participants entering the Open-label phase at study start. | 44.98 (13.25)
Gender [Number; unit: participants] — OL Baseline All Enrolled Population. Baseline Gender reported for participants entering the Open-label phase at study start.
  participants
    Female | 608 | 0 | 0 | 608
    Male | 266 | 0 | 0 | 266
Number of participants per categorical score on Clinical Global Impression-Improvement (CGI-I) scale [Number; unit: participants] — CGI-I is a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Outcome measure CGI-I results reported for DB phase; CGI-I baseline=DB baseline.
  participants
    1=very much improved | 0 | 239 | 223 | 462
    2=much improved | 0 | 36 | 49 | 85
    3=minimally improved | 0 | 1 | 0 | 1
    4=no change | 0 | 0 | 0 | 0
    5=minimally worse | 0 | 0 | 0 | 0
    6=much worse | 0 | 0 | 0 | 0
    7=very much worse | 0 | 0 | 0 | 0
Hamilton Psychiatric Scale for Depression-17 Item (HAM-D17) Total Score [Mean (Standard Deviation); unit: scores on a scale] — HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Nine items are scored on a 3 point scale (0=none/absent to 2=most severe) and 8 items are scored on a 5 point scale (0=none/absent to 4=most severe) for a maximum total score of 50; higher score indicates more depression.
  scores on a scale | NA (NA) — Outcome measure HAM-D17 results reported for DB phase; HAM-D17 baseline=DB baseline. | 4.58 (3.02) | 4.69 (2.97) | 4.64 (2.99)
Number of participants with remission based on HAM-D17 score [Number; unit: participants] — HAM-D17: standardized, clinician-administered rating scale that assesses 17 items associated with major depression (such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Nine items scored on 3 point scale (0=none/absent to 2=most severe) and 8 items scored on 5 point scale (0=none/absent to 4=most severe) for maximum total score of 50; higher score indicates more depression. Remission (Yes or No) based on HAMD-17 total score ≤7. Outcome measure HAM-D17 Remission results reported for DB phase; HAM-D17 Remission baseline=DB baseline.
  participants
    Remission=No | 0 | 46 | 52 | 98
    Remission=Yes | 0 | 230 | 220 | 450

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse Following Randomization to the Double-blind (DB) Phase: Estimated Probability (Percent) of Relapse at DB Day 185
Description: Time to relapse analyzed using log-rank test; defined as Hamilton Psychiatric Scale for Depression-17 item score ≥16 at any time during DB phase, discontinuation for unsatisfactory response or efficacy (need for additional or alternate treatment for depression, investigator decision to remove participant for efficacy reasons, or failure to return if investigator determined related to efficacy), hospitalization for depression, suicide attempt, or suicide. Participants who relapsed after DB day 185 or completed DB therapy without relapse were considered as censored on DB day 185 (study day 325).
Time Frame: Double-blind phase Baseline (Study Day 140) up to DB Day 185 (Study Day 325)
Population: All Randomized population: all participants randomly assigned to the Double-blind treatment phase of the study.
Measure: Number; unit: percent estimated probability
Groups:
- Placebo: Placebo matching DVS SR 50 mg and DVS SR 25 mg PO QD Days 141 to 147, then placebo matching DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with placebo matching DVS SR 25 mg PO QD.
- DVS SR 50 mg: DVS SR 50 mg and placebo matching DVS SR 25 mg PO QD Days 141 to 147; DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with DVS SR 25 mg PO QD.
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 276 | 272
percent estimated probability | 30.2 | 14.3
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Test type: Superiority or Other; p < 0.001, Log Rank — Significance declared if p-value ≤0.05. The estimated probability obtained via Kaplan-Meier estimate

2. Secondary Outcome: Number of Participants Per Categorical Score for Change From Baseline on Clinical Global Impression-Improvement (CGI-I) Scale
Description: CGI-I is a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale.
Time Frame: Double-blind phase Baseline (Study Day 140) up to Week 26 (Study Day 322)
Population: All Randomized population. N=number of participants with analyzable data at observation (Observed Cases).
Measure: Number; unit: participants
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 267 | 261
participants
  DB Week 1: 1=very much improved | 9 | 3
  DB Week 1: 2=much improved | 1 | 3
  DB Week 1: 3=minimally improved | 12 | 19
  DB Week 1: 4=no change | 227 | 212
  DB Week 1: 5=minimally worse | 16 | 20
  DB Week 1: 6=much worse | 2 | 3
  DB Week 1: 7=very much worse | 0 | 1
  DB Week 2: 1=very much improved | 7 | 3
  DB Week 2: 2=much improved | 5 | 6
  DB Week 2: 3=minimally improved | 15 | 24
  DB Week 2: 4=no change | 183 | 197
  DB Week 2: 5=minimally worse | 32 | 25
  DB Week 2: 6=much worse | 15 | 4
  DB Week 2: 7=very much worse | 0 | 0
  DB Week 3: 1=very much improved | 5 | 6
  DB Week 3: 2=much improved | 5 | 8
  DB Week 3: 3=minimally improved | 17 | 27
  DB Week 3: 4=no change | 169 | 185
  DB Week 3: 5=minimally worse | 45 | 24
  DB Week 3: 6=much worse | 6 | 2
  DB Week 3: 7=very much worse | 0 | 0
  DB Week 4: 1=very much improved | 5 | 8
  DB Week 4: 2=much improved | 6 | 7
  DB Week 4: 3=minimally improved | 20 | 28
  DB Week 4: 4=no change | 169 | 181
  DB Week 4: 5=minimally worse | 39 | 20
  DB Week 4: 6=much worse | 6 | 2
  DB Week 4: 7=very much worse | 1 | 1
  DB Week 6: 1=very much improved | 6 | 9
  DB Week 6: 2=much improved | 5 | 11
  DB Week 6: 3=minimally improved | 20 | 31
  DB Week 6: 4=no change | 153 | 174
  DB Week 6: 5=minimally worse | 40 | 16
  DB Week 6: 6=much worse | 14 | 6
  DB Week 6: 7=very much worse | 0 | 0
  DB Week 10: 1=very much improved | 3 | 7
  DB Week 10: 2=much improved | 4 | 9
  DB Week 10: 3=minimally improved | 19 | 28
  DB Week 10: 4=no change | 140 | 161
  DB Week 10: 5=minimally worse | 46 | 28
  DB Week 10: 6=much worse | 9 | 8
  DB Week 10: 7=very much worse | 1 | 1
  DB Week 14: 1=very much improved | 3 | 4
  DB Week 14: 2=much improved | 5 | 10
  DB Week 14: 3=minimally improved | 16 | 29
  DB Week 14: 4=no change | 124 | 159
  DB Week 14: 5=minimally worse | 49 | 25
  DB Week 14: 6=much worse | 10 | 3
  DB Week 14: 7=very much worse | 0 | 0
  DB Week 18: 1=very much improved | 6 | 7
  DB Week 18: 2=much improved | 6 | 6
  DB Week 18: 3=minimally improved | 12 | 28
  DB Week 18: 4=no change | 117 | 151
  DB Week 18: 5=minimally worse | 39 | 24
  DB Week 18: 6=much worse | 12 | 6
  DB Week 18: 7=very much worse | 0 | 1
  DB Week 22: 1=very much improved | 7 | 8
  DB Week 22: 2=much improved | 4 | 6
  DB Week 22: 3=minimally improved | 13 | 29
  DB Week 22: 4=no change | 116 | 139
  DB Week 22: 5=minimally worse | 30 | 28
  DB Week 22: 6=much worse | 13 | 5
  DB Week 22: 7=very much worse | 1 | 0
  DB Week 26: 1=very much improved | 7 | 9
  DB Week 26: 2=much improved | 7 | 10
  DB Week 26: 3=minimally improved | 13 | 29
  DB Week 26: 4=no change | 105 | 135
  DB Week 26: 5=minimally worse | 31 | 22
  DB Week 26: 6=much worse | 10 | 5
  DB Week 26: 7=very much worse | 1 | 0

3. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Illness [CGI-S] Score in the Double-blind Phase
Description: CGI-S is a 7-point clinician rated scale to assess severity of participant's current illness state; range of 1 (normal - not ill at all) to 7 (among the most extremely ill). Higher score = more affected. Change from baseline mean=adjusted mean change calculated using mixed-effects model for repeated measures (MMRM).
Time Frame: Double-blind phase Baseline (Study Day 140) up to Week 26 (Study Day 322)
Population: All Randomized population. N=number of participants with analyzable data at observation.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 267 | 261
scores on a scale
  Change from Baseline at DB Week 1 | 0.03 (0.03) | 0.03 (0.03)
  Change from Baseline at DB Week 2 | 0.18 (0.04) | 0.09 (0.04)
  Change from Baseline at DB Week 3 | 0.21 (0.04) | 0.07 (0.04)
  Change from Baseline at DB Week 4 | 0.23 (0.05) | 0.06 (0.05)
  Change from Baseline at DB Week 6 | 0.32 (0.05) | 0.06 (0.05)
  Change from Baseline at DB Week 10 | 0.39 (0.06) | 0.11 (0.06)
  Change from Baseline at DB Week 14 | 0.38 (0.05) | 0.05 (0.05)
  Change from Baseline at DB Week 18 | 0.42 (0.06) | 0.09 (0.06)
  Change from Baseline at DB Week 22 | 0.56 (0.07) | 0.13 (0.07)
  Change from Baseline at DB Week 26 | 0.53 (0.06) | 0.09 (0.06)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 1; Test type: Superiority or Other; p = 0.9627, Mixed Models Analysis — P-value obtained from mixed model: change from baseline = baseline + site + treatment + visit + treatment*visit with "Unstructured" covariance structure; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.09 to 0.08]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 2; Test type: Superiority or Other; p = 0.1046, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.02 to 0.21]
Statistical Analysis 3: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 3; Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.02 to 0.25]
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 4; Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.05 to 0.29]
Statistical Analysis 5: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 6; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.11 to 0.39]
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 10; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.12 to 0.43]
Statistical Analysis 7: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.33, 95% CI 2-sided [0.19 to 0.47]
Statistical Analysis 8: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 18; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.33, 95% CI 2-sided [0.17 to 0.49]
Statistical Analysis 9: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 22; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.43, 95% CI 2-sided [0.25 to 0.62]
Statistical Analysis 10: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.44, 95% CI 2-sided [0.28 to 0.61]

4. Secondary Outcome: Change From Baseline in Hamilton Psychiatric Scale for Depression-17 Item (HAM-D17) Score in the Double-blind Phase
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Nine items are scored on a 3 point scale (0=none/absent to 2=most severe) and 8 items are scored on a 5 point scale (0=none/absent to 4=most severe) for a maximum total score of 50; higher score indicates more depression. Change from baseline mean=adjusted mean change calculated using MMRM.
Time Frame: Double-blind phase Baseline (Study Day 140) up to Week 26 (Study Day 322)
Population: All Randomized population. N=number of participants with analyzable data at observation.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 267 | 261
scores on a scale
  Change from Baseline at DB Week 1 | 0.28 (0.17) | 0.25 (0.17)
  Change from Baseline at DB Week 2 | 1.40 (0.24) | 0.53 (0.24)
  Change from Baseline at DB Week 3 | 1.32 (0.22) | 0.45 (0.23)
  Change from Baseline at DB Week 4 | 1.50 (0.24) | 0.11 (0.24)
  Change from Baseline at DB Week 6 | 1.94 (0.28) | 0.31 (0.28)
  Change from Baseline at DB Week 10 | 2.37 (0.32) | 0.69 (0.31)
  Change from Baseline at DB Week 14 | 2.66 (0.30) | 0.62 (0.30)
  Change from Baseline at DB Week 18 | 2.51 (0.33) | 0.56 (0.32)
  Change from Baseline at DB Week 22 | 3.22 (0.37) | 0.92 (0.36)
  Change from Baseline at DB Week 26 | 3.12 (0.36) | 0.77 (0.34)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 1; Test type: Superiority or Other; p = 0.8853, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.41 to 0.47]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 2; Test type: Superiority or Other; p = 0.0081, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.88, 95% CI 2-sided [0.23 to 1.52]
Statistical Analysis 3: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 3; Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.88, 95% CI 2-sided [0.28 to 1.47]
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 4; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.39, 95% CI 2-sided [0.76 to 2.03]
Statistical Analysis 5: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 6; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.63, 95% CI 2-sided [0.86 to 2.39]
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 10; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.68, 95% CI 2-sided [0.83 to 2.54]
Statistical Analysis 7: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 2.04, 95% CI 2-sided [1.23 to 2.86]
Statistical Analysis 8: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 18; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.95, 95% CI 2-sided [1.06 to 2.84]
Statistical Analysis 9: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 22; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 2.30, 95% CI 2-sided [1.31 to 3.30]
Statistical Analysis 10: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 2.35, 95% CI 2-sided [1.39 to 3.32]

5. Secondary Outcome: Change From Baseline in Hamilton Psychiatric Scale for Depression-6 Item (HAM-D6) Score in the Double-blind Phase
Description: HAM-D6 is a standardized, clinician-administered rating scale is a subset of the HAM-D17 that assesses 6 items associated with major depression. The scale uses HAM-D17 items 1, 2, 7, 8, 10 and 13. Item 13 is scored 0 to 2 (0=none/absent to 2=most severe) and all others are scored 0 to 4 (0=none/absent to 4=most severe). Total score ranges from 0 to 22; higher score indicates more depression. Change from baseline mean=adjusted mean change calculated using MMRM.
Time Frame: Double-blind phase Baseline (Study Day 140) up to Week 26 (Study Day 322)
Population: All Randomized population. N=number of participants with analyzable data at observation.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 267 | 261
scores on a scale
  Change from baseline at DB Week1 | 0.03 (0.10) | 0.01 (0.10)
  Change from baseline at DB Week 2 | 0.66 (0.14) | 0.13 (0.14)
  Change from baseline at DB Week 3 | 0.72 (0.14) | 0.14 (0.14)
  Change from baseline at DB Week 4 | 0.92 (0.15) | 0.03 (0.15)
  Change from baseline at DB Week 6 | 1.04 (0.17) | 0.16 (0.16)
  Change from baseline at DB Week 10 | 1.41 (0.19) | 0.33 (0.18)
  Change from baseline at DB Week 14 | 1.47 (0.17) | 0.34 (0.17)
  Change from baseline at DB Week 18 | 1.51 (0.20) | 0.21 (0.19)
  Change from baseline at DB Week 22 | 1.68 (0.20) | 0.45 (0.19)
  Change from baseline at DB Week 26 | 1.53 (0.20) | 0.26 (0.19)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 1; Test type: Superiority or Other; p = 0.9142, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.24 to 0.27]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 2; Test type: Superiority or Other; p = 0.0069, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.53, 95% CI 2-sided [0.15 to 0.91]
Statistical Analysis 3: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 3; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.58, 95% CI 2-sided [0.21 to 0.95]
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 4; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.89, 95% CI 2-sided [0.49 to 1.28]
Statistical Analysis 5: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 6; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 0.88, 95% CI 2-sided [0.43 to 1.32]
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 10; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.58 to 1.58]
Statistical Analysis 7: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.12, 95% CI 2-sided [0.66 to 1.58]
Statistical Analysis 8: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 18; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.30, 95% CI 2-sided [0.76 to 1.83]
Statistical Analysis 9: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 22; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.23, 95% CI 2-sided [0.70 to 1.76]
Statistical Analysis 10: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.27, 95% CI 2-sided [0.75 to 1.79]

6. Secondary Outcome: Number of Participants With Remission Based on Hamilton Psychiatric Scale for Depression-17 Item (HAM-D17) Score at Double-blind Phase Week 26
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Nine items are scored on a 3 point scale (0=none/absent to 2=most severe) and 8 items are scored on a 5 point scale (0=none/absent to 4=most severe) for a maximum total score of 50; higher score indicates more depression. Remission defined as HAM-D17 total score ≤7.
Time Frame: Double-blind phase Week 26 (Study Day 322)
Population: All Randomized population. N=number of participants with analyzable data at observation based on Last Observation Carried Forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 273 | 270
participants | 148 | 201
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Wald 95% CI for adjusted odds ratio; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Obtained from logistic regression analysis using Remission (Yes/No) at each time point as a response variable; logistic model with treatment and sites as factors and baseline HAM-D17 total score as covariate; Adjusted odds ratio = 2.85, 95% CI 2-sided [1.93 to 4.20]

7. Secondary Outcome: Change From Baseline of Double-blind Phase in World Health Organization (Five-Item) Well-Being Index
Description: WHO-5 evaluates positive psychological well-being during the past 2 weeks and consists of 5 questions (felt cheerful, in good spirits; felt calm, relaxed; felt active, vigorous; woke up fresh, rested; and daily life filled with things that are interesting) each rated on a 6-point Likert scale from 0 (not present) to 5 (constantly present). Total raw score ranged from 0 (worst possible quality of life) to 25 (best possible quality of life). Change from baseline mean=adjusted mean change calculated using MMRM.
Time Frame: Double-blind phase Baseline (Study Day 140), Week 14 (Study Day 238), Week 26 (Study Day 322)
Population: All Randomized population. N=number of participants with analyzable data at observation.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 265 | 261
scores on a scale
  Change from baseline at DB Week 14 | -2.51 (0.35) | -0.38 (2.36)
  Change from baseline at DB Week 26 | -2.36 (0.38) | -0.04 (0.37)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value obtained from mixed model: change from baseline = baseline + treatment + visit + treatment*visit with "Unstructured" covariance structure; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-3.03 to -1.24]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = -2.32, 95% CI 2-sided [-3.29 to -1.34]

8. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) Score in the Double-blind Phase
Description: WPAI is a 6 question participant rated questionnaire to determine the degree to which depression affected work productivity while at work and affected activities outside of work. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combined absenteeism and presenteeism and percentage of impairment in activities performed outside of work. Scores scaled as 0 (not affected/no impairment) to 10 (completely affected/impaired). Higher score indicated greater impairment and less productivity.
Time Frame: Double-blind phase Baseline (Study Day 140), Week 14 (Study Day 238), Week 26 (Study Day 322)
Population: All Randomized population. Change from baseline (Bsl) mean=adjusted mean change calculated using MMRM.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | DVS SR 50 mg
Number analyzed (Participants) | 265 | 261
scores on a scale
  Change from Bsl at DB Week 14: Absenteeism | 1.64 (1.72) | 0.62 (1.87)
  Change from Bsl at DB Week 14: Presenteeism | 9.35 (2.30) | 2.44 (2.55)
  Change from Bsl DB Week 14: Work productivity loss | 9.66 (2.48) | 2.19 (2.75)
  Change from Bsl at DB Week 14: Activity impairment | 11.02 (1.62) | 3.45 (1.66)
  Change from Bsl at DB Week 26: Absenteeism | 0.43 (2.05) | 0.77 (2.08)
  Change from Bsl at DB Week 26: Presenteeism | 7.75 (2.35) | -0.49 (2.41)
  Change from Bsl DB Week 26: Work productivity loss | 8.47 (2.56) | -0.00 (2.63)
  Change from Bsl at DB Week 26: Activity impairment | 9.67 (1.75) | 2.05 (1.69)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14 Absenteeism; Test type: Superiority or Other; p = 0.6772, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.02, 95% CI 2-sided [-3.82 to 5.87]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26 Absenteeism; Test type: Superiority or Other; p = 0.9059, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-5.91 to 5.24]
Statistical Analysis 3: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14 Presenteeism; Test type: Superiority or Other; p = 0.0414, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 6.91, 95% CI 2-sided [0.27 to 13.55]
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26 Presenteeism; Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 8.24, 95% CI 2-sided [1.77 to 14.71]
Statistical Analysis 5: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14 Work Productivity Loss; Test type: Superiority or Other; p = 0.0402, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 7.48, 95% CI 2-sided [0.34 to 14.61]
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26 Work Productivity Loss; Test type: Superiority or Other; p = 0.0187, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 8.48, 95% CI 2-sided [1.43 to 15.53]
Statistical Analysis 7: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 14 Activity Impairment; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 7.57, 95% CI 2-sided [3.33 to 11.80]
Statistical Analysis 8: Comparison: Placebo vs DVS SR 50 mg; Adjusted difference from placebo: Week 26 Activity Impairment; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 7.62, 95% CI 2-sided [3.14 to 12.10]

ADVERSE EVENTS:
Time Frame: Events collected from the time informed consent in Open-Label phase (OL) through 15 days after last dose or up to study day 336.
Description: Same event may appear as both an AE and SAE, however, are presented as distinct events; may be categorized as SAE in 1 subject and as non-SAE in another, or 1 subject may have experienced both an SAE and non-SAE during study. Participants are counted multiple times: transition from OL Response to OL Stability phase; then as randomized to DB phase.
Groups:
- DVS SR 50 mg (Open-label Response Phase): DVS SR 50 mg PO QD for 8 weeks.
- DVS SR 50 mg (Open Label Stability Phase): DVS SR 50 mg PO QD; Responders at week 8 entered a 12-week stability phase.
- DVS SR 50 mg (Open Label Taper / OL Post Study Follow Up): Participants who concluded DVS SR 50 mg open-label study or discontinued treatment at any time in OLR or OLS could have entered the taper phase and received DVS SR 25 mg PO QD for a 7-day period of taper treatment. N=number of participants with OL Taper or OL Post Study Follow Up emergent events who did not enter the DB Phase and concluded or discontinued with or without taper treatment.
- Placebo (Double-blind Phase): Placebo matching DVS SR 50 mg and DVS SR 25 mg PO QD Days 141 to 147, then placebo matching DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with placebo matching DVS SR 25 mg PO QD.
- DVS SR 50 mg (Double-blind Phase): DVS SR 50 mg and placebo matching DVS SR 25 mg PO QD Days 141 to 147; DVS SR 50 mg PO QD Days 148 to 322 followed by 7-day taper period with DVS SR 25 mg PO QD.
- Placebo (DB Taper / DB Post Study Follow Up): Participants who concluded or discontinued placebo during the DB phase could have entered the taper phase and received placebo matching DVS SR 25 mg for a 7-day period of taper treatment. N=number of participants with DB Taper or DB Post Study Follow Up emergent events who concluded or discontinued with or without taper treatment.
- DVS SR 50 mg (DB Taper / DB Post Study Follow Up): Participants who concluded or discontinued DVS SR 50 mg during the DB phase could have entered the taper phase and received DVS SR 25 mg for a 7-day period of taper treatment. N=number of participants with DB Taper or DB Post Study Follow Up emergent events who concluded or discontinued with or without taper treatment.
Arm/Group | DVS SR 50 mg (Open-label Response Phase) | DVS SR 50 mg (Open Label Stability Phase) | DVS SR 50 mg (Open Label Taper / OL Post Study Follow Up) | Placebo (Double-blind Phase) | DVS SR 50 mg (Double-blind Phase) | Placebo (DB Taper / DB Post Study Follow Up) | DVS SR 50 mg (DB Taper / DB Post Study Follow Up)
Serious Adverse Events (participants affected / at risk) | 9/874 | 6/659 | 4/326 | 7/276 | 8/272 | 1/276 | 1/272
Other Adverse Events (participants affected / at risk) | 609/874 | 36/659 | 8/326 | 81/276 | 55/272 | 14/276 | 23/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 mg (Open-label Response Phase) (N=874) | DVS SR 50 mg (Open Label Stability Phase) (N=659) | DVS SR 50 mg (Open Label Taper / OL Post Study Follow Up) (N=326) | Placebo (Double-blind Phase) (N=276) | DVS SR 50 mg (Double-blind Phase) (N=272) | Placebo (DB Taper / DB Post Study Follow Up) (N=276) | DVS SR 50 mg (DB Taper / DB Post Study Follow Up) (N=272)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Self injurious behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Outcome: Death
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intrauterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 mg (Open-label Response Phase) (N=874) | DVS SR 50 mg (Open Label Stability Phase) (N=659) | DVS SR 50 mg (Open Label Taper / OL Post Study Follow Up) (N=326) | Placebo (Double-blind Phase) (N=276) | DVS SR 50 mg (Double-blind Phase) (N=272) | Placebo (DB Taper / DB Post Study Follow Up) (N=276) | DVS SR 50 mg (DB Taper / DB Post Study Follow Up) (N=272)
Constipation (Gastrointestinal disorders) | 51 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 44 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 104 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 184 | 0 | 0 | 0 | 0 | 1 | 7
Dizziness (Nervous system disorders) | 62 | 0 | 0 | 29 | 13 | 1 | 13
Headache (Nervous system disorders) | 160 | 36 | 8 | 35 | 34 | 4 | 7
Somnolence (Nervous system disorders) | 45 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 44 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 50 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 17 | 8 | 9 | 3

LIMITATIONS AND CAVEATS:
P-value from the primary analysis is different from the one testing equality of relapse rates on Double-blind day 185. Estimated percentages were provided as representative descriptive measures. Medians were not estimable due to low relapse rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.